CLINICAL TRIAL: NCT02910791
Title: The Role of Bacterial Toxins in Human Skin Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Donald Leung, MD, PhD, Principal Investigator, National Jewish Health
Other Study IDs: HS-3008
Record Dates: First submitted 2016-09-13; First posted 2016-09-22 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- atopic dermatitis: up to 40 subjects with atopic dermatitis will be enrolled into study.
- psoriasis: up to 20 subjects with psoriasis will be enrolled into study.
- people without skin conditions: Up to 40 subjects without skin conditions will be enrolled into study.

SUMMARY:
Atopic dermatitis and psoriasis are two skin diseases often associated with bacterial infections and inflammation. Studies indicate that skin cells from these patients may have some changes that make these patients more susceptible to bacterial infections. Inflammatory environment may have an effect on the function of skin cells.

The purpose of this study is to learn more about skin cells (keratinocytes and fibroblasts) and how they regulate skin barrier function. To study this we need to establish skin cells that can be grown in the laboratory. We will use small skin biopsies from patients with atopic dermatitis, psoriasis and healthy people as a source of these cells. Since these skin cells have a limited lifetime when grown in laboratory as part of the project we would like to modify them, which allows them to grow for long time in the research laboratory. Some of the collected skin biopsies and isolated skin cells will be used to examine what gene products they make.

DETAILED DESCRIPTION:
Visit 1 (if needed). Study subjects will be asked to read and sign the informed consent. At that time the study inclusion and exclusion criteria for the study will be reviewed. Subject will be given instructions to stop taking certain medications for 7 days prior to the next study visit. Alternatively, if Visit 1 will be done over the phone, subjects may be contacted via phone using a phone script to provide instructions for stopping these medications. In this case, the informed consent will be obtained by the subject at visit 2 prior to any study procedures being done.

If the subject takes occasional Aspirin (not taken daily), it will need to be withheld for seven days prior to visit 2.

If the subject takes oral antihistamines, it will need to be withheld for seven days prior to the subject's first appointment.

If the subject takes oral antibiotics, inform the subject the appointment can be scheduled seven days after their last dose of antibiotic has been taken.

If the subject takes topical medications including (but not restricted to), cyclosporine, Elidel, Protopic, topical corticosteroids and topical antibiotics, it will need to be withheld seven days prior to the subject's first appointment.

If the subject takes any of the following medications, they are not eligible for enrollment:

Oral corticosteroids Any systemic immunosuppressive or immunomodulary medication in the last 28 days.

Patients who have received immunotherapy in the past year. Patients using anxiolytics or antidepressants Antiviral therapies Anticoagulants Allergic to lidocaine Daily Aspirin

Visit 2: Will occur approximately 7 days following the screening visit or the phone call. If the subject was contacted via phone, he/she will be review and sign the informed consent form during this visit. The following procedures will be performed.

Urine Pregnancy Test: All female can be pregnant or become pregnant during the study. The urine pregnancy test will be administered to all women of child bearing potential. If the test will be positive, the participation in the study will be terminated.

Skin Biopsies: The skin biopsies will involve taking a small piece of skin (4 biopsies 2mm in diameter) generally obtained from the arms or legs, the face is excluded from skin biopsy. The area will be cleaned and numbed with a local anesthetic. Biopsies will be collected from non-lesion skin and acute lesions. The wound will not require a stitch and should be healed within two weeks. The biopsy site needs to be kept sterile and this will require that the area not get wet. The skin biopsies will be performed by one of the physician investigators or nurse practitioners. The subject will be given the name and phone number of a nurse and told to call if there are any problems. The subject will be given instructions on how to care for the biopsy site.

Venipuncture: 7.5 mL of blood will be removed by putting a needle into a vein. The procedure will be performed by a physician investigator or a nurse in the CTRC. The subject will be given the name and phone number of a nurse and told to call if there are any problems. There will not be any follow-up for venipuncture procedures.

DNA testing: Additional 7.5 ml of blood will be obtained for genetic testing of filaggrin gene polymorphisms (performed by ADx lab at NJH).

Skin cultures: Skin is rubbed with a cotton swab then cells are placed in a special culture medium tube for identification of bacteria wabs will be tested for presence of S. aureus by culture and PCR.

Tape Stripping. Adhesive skin sampling discs will be firmly pressed against the skin in a hairless location (not the face) followed by lifting it free of the skin. Skin tapes will be collected from non-lesion skin and acute skin lesions. This will be repeated up to 40 times. These discs will then be used to evaluate RNA, lipids and proteins in the upper layers of skin. With every 5 tape strips collected from one lesion and one non-lesion area skin barrier assessment will be preformed.

Skin Barrier Assessment. Skin serves as the first barrier against allergens, viruses, and bacteria that may aggravate your skin disease. A small device will be used to measure the quantity of water that passes from inside the body through the skin to the surrounding atmosphere via diffusion and evaporation process. Additionally, the device will measure skin pH, which is also associated with changes in the skin barrier.

Sweat Test. We will measure chemicals in patients' sweat, such as salt, which is known as a sweat test. To collect the sweat, a sticky pad will be attached to the skin on patients' arm for 5 minutes. A gel containing a medicine called pilocarpine is put on the pads and causes the sweat glands to produce more sweat. The pads are then removed and replaced by a disc to collect sweat for about 30 minutes.

Sebum Collection. Skin surface will be cleaned with alcohol wipes. After allowing skin surface to dry sebum collecting tape will be applied to the skin surface. The tape will be held on the skin surface for one hour. The tape will then be used to evaluate skin sebum production.

Optional Visits: The research team may ask the subject to return every 6 weeks and participate in additional skin biopsies, tape strips and blood draws (not to exceed 6.5 tablespoons (100 ml)). The subject may choose to participate in some or all optional visits not to exceed 6 additional blood draws, tape strips and/or biopsies in one year.

ELIGIBILITY:
Inclusion Criteria:

* If subjects takes occasional Aspirin (not taken daily), it will need to be withheld for seven days prior to Visit 2.
* If subjects takes oral antihistamines, it will need to be withheld for seven days prior to the subject's first appointment
* If subjects takes topical medications including (but not restricted to), cyclosporine, Elidel, Protopic, topical corticosteroids and topical antibiotics, it will need to withheld seven days prior to the subject's first appointment.

Exclusion Criteria:

* Women can not be pregnant or become pregnant during the study
* Oral corticosteroids:

  * Any systemic immunosuppressive or immunomodulatory medication in the last 28 days.
  * Patients who have received immunotherapy in the past year.
  * Patients using anxiolytics or antidepressants
  * Antiviral therapies
  * Anticoagulants
  * Allergic to lidocaine
  * Daily Aspirin use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of adults (18-65 years old) with AD, psoriasis or healthy controls with no history of chronic skin diseases and atopy. Recruitment will aim for up to 40 subjects with AD, up to 20 subjects with psoriasis, and up to 40 healthy normal controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To determine the molecular mechanisms by which cytokines in atopic dermatitis skin alters differentiation of skin keratinocytes | one year

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided